CLINICAL TRIAL: NCT05550493
Title: Preliminary Efficacy of a Digital Therapeutics Smartphone Application for Methamphetamine Use Disorder
Brief Title: Digital Therapeutics Smartphone Application for Methamphetamine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Collaborators: Huangshui Township Municipal Government, Shuangliu District, Chengdu, Sichuang (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Feidao
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Methamphetamine Abuse
MeSH Terms: interventions — Cognitive Behavioral Therapy; Counseling; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Therapeutics (Experimental): The DTx group was asked to download and install a smartphone application (WonderLab Harbor) that incorporated Internet-based Cognitive Behavioral Therapy (ICBT), Approach Bias Modification (ApBM), cognitive function training, and Contingency Management (CM). During the 8-week treatment program, the participants in the DTx group were instructed to complete ICBT, cognitive trainings, and ApBM trainings. Reward points (which can be redeemed for cellphone plan credit) were rewarded following completing each task as part of the positive reinforcement following CM principles.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Approach Bias Modification; Behavioral: Cognitive Training
- Treatment as Usual (Active Comparator): Upon enrollment, TAU participants were informed that they would receive weekly counseling sessions from a social worker for eight weeks. The counseling covered topics including work, family, stress management, and drug craving suppression.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The cognitive behavioral therapy program consisted of eight interactive sessions, each requiring approximately 15 minutes to complete. Each ICBT session includes interactive multimedia modules (videos, pictures, and texts), the contents of which were based on the community reinforcement approach. The ICBT sessions covered the following topics: (1) introduction to digital therapeutics and CBT, (2) recognizing the triggers of craving, (3) coping with craving, (4) refusing skills/assertiveness, (5) problem-solving skills, (6) changing thoughts about drugs, (7) seemingly irrelevant decisions, and (8) HIV risks and prevention.
  Arms: Digital Therapeutics
Behavioral: Counseling — Counseling provided by social workers and psychotherapists on topics including work, family, stress management, and drug craving suppression.
  Arms: Treatment as Usual
Behavioral: Approach Bias Modification — In an ApBM session, users were instructed to swipe upward (downward) when they saw portrait (landscape) format images. A shrinking (growing) animation comes after swiping upward (downward) to simulate the visual effect of moving away (moving towards). The images were related to methamphetamine usage (methamphetamine crystals, powders, and paraphernalia) or healthy lifestyles (wealth, sports, gourmet, family activities, etc.). Each ApBM session was composed of presenting each one of the healthy lifestyle (methamphetamine) cues 12 times in landscape (portrait) and once in portrait (landscape).
  Arms: Digital Therapeutics
Behavioral: Cognitive Training — The DTx application incorporated a game-based cognitive function training module for improving working memory. In this game, a matrix of squares is displayed at the center of the screen. Between 3 and 5 target symbols are randomly placed in the matrix and displayed for 2 seconds. Next, the symbols disappear, and the matrix randomly rotates. The participants were asked to click the correct locations of the target symbols within the prescribed time limit. The game becomes more difficult as the size of the matrix, the number of target symbols, and the complexity of the matrix rotation change at each level. Each cognitive function training session lasted between 3 and 5 minutes.
  Arms: Digital Therapeutics

SUMMARY:
One hundred participants were recruited and randomized into a digital therapeutics (DTx) group (n=52) and a treatment as usual (TAU) group (n=48). The DTx group used a smartphone application to deliver cognitive behavioral therapy, approach bias modification, cognitive training, and contingency management for eight weeks. The TAU group received counseling from social workers and psychoterapists. Cue-induced craving, cognitive functions, PHQ-9, and GAD-7 were measured at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* currently undergoing community-based rehabilitation were recruited voluntarily from four community
* meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for methamphetamine dependence.

Exclusion Criteria:

* could not fluently operate an Android or an iOS smartphone
* having mental health conditions other than MUD

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Cue induced craving for methamphetamine | baseline, pre-intervention
  The cue-induced craving was assessed by showing the participants images related to methamphetamine (methamphetamine crystals, powders, and paraphernalia) on a smartphone and asking them to rate their cravings on a 0-10 visual analog scale (0 being least craved and 10 being most craved).
Cue induced craving for methamphetamine | immediately after the intervetion
  The cue-induced craving was assessed by showing the participants images related to methamphetamine (methamphetamine crystals, powders, and paraphernalia) on a smartphone and asking them to rate their cravings on a 0-10 visual analog scale (0 being least craved and 10 being most craved).
Cognitive Function Score | baseline, pre-intervention
  We use the Meaningless Figure Recognition Test (MFRT) to assess the cognitive function score. This test has eight blocks, and each block has two phases. In the first phase, the participant is presented with a series of meaningless figures one by one for three seconds. The participants were asked to memorize these figures. In the second phase, the previously presented meaningless figures and the same number of the novel meaningless figures are presented on one screen in random order. The participants were asked to recall their memory and click all the previously presented figures within 15 seconds. The correct rate of clicks is used for measuring the cognitive function scores.
Cognitive Function Score | immediately after the intervetion
  We use the Meaningless Figure Recognition Test (MFRT) to assess the cognitive function score. This test has eight blocks, and each block has two phases. In the first phase, the participant is presented with a series of meaningless figures one by one for three seconds. The participants were asked to memorize these figures. In the second phase, the previously presented meaningless figures and the same number of the novel meaningless figures are presented on one screen in random order. The participants were asked to recall their memory and click all the previously presented figures within 15 seconds. The correct rate of clicks is used for measuring the cognitive function scores.

SECONDARY OUTCOMES:
PHQ-9 | baseline, pre-intervention
  Patient Health Questionaire-9 administered on a smartphone
PHQ-9 | immediately after the intervetion
  Patient Health Questionaire-9 administered on a smartphone
GAD-7 | baseline, pre-intervention
  Generalized Anxiety Disorder 7-item administered on a smartphone
GAD-7 | immediately after the intervetion
  Generalized Anxiety Disorder 7-item administered on a smartphone

CONTACTS AND LOCATIONS:
Locations (1):
- Huangshui Township Municipal Government, Chengdu, Sichuang, China

IPD SHARING:
Plan to Share IPD: No